CLINICAL TRIAL: NCT01347905
Title: Changes in Iron Absorption and Availability Before and After Weight Loss in Obese Pre-menopausal Women and Men.
Status: Completed | Type: Observational
Sponsor: Wageningen University (Other)
Collaborators: Universidad de Monterrey (Other); Mexican National Institute of Public Health (Other Government); Swiss Federal Institute of Technology (Other); Unilever R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: Iron absorption and obesity
Record Dates: First submitted 2011-05-03; First posted 2011-05-05 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood and serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Obese women and men: Obese women and men undergoing restrictive bariatric surgery. Iron absorption will be estimated using stable-isotope techniques where incorporation of 57Fe and 58Fe into erythrocytes is measured 14 days after administration. This procedure will be performed at baseline (6 weeks post-surgery) and at the end of the study (6-7 months post baseline).
  Interventions: Other: Stable-isotope techniques

INTERVENTIONS:
Other: Stable-isotope techniques — Iron absorption will be estimated using stable-isotope techniques where incorporation of 57Fe and 58Fe into erythrocytes is measured 14 days after administration. The subjects will provide an initial blood sample (20ml) and then receive a test drink, containing 6 mg of 57Fe labeled ferrous sulphate. One hour later, 2 ml of an aqueous solution containing 100 μg 58Fe, as iron citrate in 250cc of normal saline will be infused over 50 min. Post infusion a 4ml blood sample will be taken. This procedure will be performed at baseline (6 weeks post-surgery) and at the end of the study (6-7 months post baseline).
  Other Names: 57Fe ferrous sulphate; 58Fe iron citrate

SUMMARY:
The objective of this study is to investigate if weight loss, in particular due to adipose tissue loss, in obese patients will reverse the obesity-related reduction of iron absorption, and if this is due to a decrease in hepcidin concentrations. Additionally, the investigators will investigate changes in iron incorporation into erythrocytes due to a reduction of iron sequestration by the adipose tissue and reticuloendothelial system. The investigators expect that by decreasing adiposity, circulating hepcidin levels will decrease, iron absorption and incorporation into erythrocytes will increase and as a result iron status will be improved.

DETAILED DESCRIPTION:
Until now adiposity has been associated with low iron status and with higher hepcidin levels. Moreover, weight loss and thereby loss of fat mass, has been associated with decreased hepcidin levels and improved iron status. However, until now no direct measures of iron absorption or incorporation into erythrocytes have been assessed before and after losing weight/fat mass.

We hypothesize that:

* body fat loss in obese women and men will improve iron absorption, corrected for iron status, from a labeled test meal measured by using a stable isotopes technique by on average 30%.
* body fat loss in obese women and men will decrease the related inflammatory state.
* greater subclinical inflammation in obese women and men will be correlated with a decreased incorporation of iron into erythrocytes, and that this will improve after loss of body fat.

The study is a prospective cohort in which iron bioavailability will be assessed in obese women and men before and after weight loss and associated loss of body fat over a period of 6 months.

Iron absorption will be estimated using stable-isotope techniques where incorporation of 57Fe and 58Fe into erythrocytes is measured 14 days after administration. Preparation of isotopically labelled iron will be done at the Laboratory of Human Nutrition of the Swiss Federal Institute of Technology Zurich (ETH Zürich).

A baseline venous blood sample will be drawn 6-8 weeks after the surgery when surgery-related inflammation has been resolved. The subjects will receive a test drink, containing 6 mg of 57Fe labelled ferrous sulphate. One hour later, 2 ml of an aqueous solution containing 100 μg 58Fe as iron citrate in 250 cc of normal saline will be infused over 50 min. This infusion protocol has been used safely and successfully to examine iron metabolism in both adults and infants. Fourteen days later, a second venous blood sample will be drawn. This procedure will be performed at baseline (6-8 weeks post-surgery) and at the end of the study (6 months post baseline).

Our study could provide important information to establish the mechanism by which obesity-mediated inflammation could induce iron deficiency. This will be the first human trial that will evaluate if the obesity-related reduction of iron absorption is reversible in a context where obesity and iron deficiency are both highly prevalent.

ELIGIBILITY:
Inclusion Criteria:

* Women and men
* aged 18 to 50 years
* Premenopausal (had no absence of menstrual cycle in the past 12 months)
* BMI ≥35<45
* Indication for laparoscopic Sleeve Gastrectomy (LSG) or Laparoscopic Adjustable Gastric Band (LAGB).

Subjects are eligible for this surgery if they:

1. have BMI ≥35<45 and one of the following two conditions:

   * Medical, physical or psychosocial problems associated with their obesity.
   * A history of prolonged attempts at weight loss by other means.
2. have been adequately informed and understood and accepted the potential -- risks and benefits of the procedure, and expressed a commitment to follow the rules regarding eating and exercise permanently after the procedure.

   * No postoperative complications after the surgery
   * Apparently healthy: no significant medical conditions that could influence iron or inflammatory status other than obesity (i.e., cancer, HIV/AIDS, inflammatory bowel disease, gastrointestinal bleeding, and rheumatoid arthritis, renal disease or hemochromatosis) (judged by study physician).
   * No use of medication which interferes with study measurements (as judged by the study physician)
   * Willing to not change their intake of dietary iron and not take additional iron supplements, other than provided by the study team, between baseline and study end.
   * Not being pregnant during the study period or in the six months prior to the study and not planning to become pregnant until at least 3 months after the last study visit.
   * Non-lactating in the 6 weeks prior to the study and for the duration of the study
   * No reported weight loss ≥ 10 % of bodyweight during a period of six months before pre-surgery examination.
   * No full or partial hysterectomy in the past 3 months
   * Informed consent signed
   * Agreeing to be informed about medically relevant personal test-results by a physician.
   * Agreeing to be informed about medically relevant personal test-results by a physician.
   * No reported participation in night shift work two weeks prior to pre-study investigation and during the study. Night work is defined as working between midnight and 6.00 AM.
   * Consumption of =< 14 alcoholic drinks in a typical week
   * Strenuous exercise =< 10 hours per week

Exclusion Criteria:

* Reported excessive blood loss at surgery (> 500 ml) and/or moderate/severe anemic (Hb < 100 g/L)
* Complications during restrictive bariatric surgery defined as either:
* Surgery duration of > 3 hours
* Blood loss of > 500 ml
* Perforation of the gastrointestinal tract
* Inability to adjust lapband
* Women and men with diagnosed abnormalities in iron metabolism (diagnosed from routine pre-surgery blood sample)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Obese, premenopausal women and men aged 18 to 50 years after having undergone restrictive bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2011-02; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption before and after weight loss, based on 57Fe and 58Fe isotope concentrations in erythrocytes. | 6 months

SECONDARY OUTCOMES:
Iron status and regulatory markers (Hb, serum ferritin, transferrin receptor, hepcidin),(pro)inflammatory markers (CRP, AGP, TNF-α, IL-6, leptin), blood volume, body composition (DXA). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Zimmermann, MD PHD, Study Director — Wageningen University
Locations (1):
- Universidad de Monterrey (UDEM) División de Ciencias de la Salud, San Pedro Garza García, Nuevo León, Mexico

REFERENCES:
- [Derived] Cepeda-Lopez AC, Allende-Labastida J, Melse-Boonstra A, Osendarp SJ, Herter-Aeberli I, Moretti D, Rodriguez-Lastra R, Gonzalez-Salazar F, Villalpando S, Zimmermann MB. The effects of fat loss after bariatric surgery on inflammation, serum hepcidin, and iron absorption: a prospective 6-mo iron stable isotope study. Am J Clin Nutr. 2016 Oct;104(4):1030-1038. doi: 10.3945/ajcn.115.115592. Epub 2016 Aug 24. PMID 27557657
- See also: Does obesity increase risk for iron deficiency? A review of the literature and the potential mechanisms. — http://www.ncbi.nlm.nih.gov/pubmed/21462109
- See also: Sharply higher rates of iron deficiency in obese Mexican women and children are predicted by obesity-related inflammation rather than by differences in dietary iron intake. — http://www.ncbi.nlm.nih.gov/pubmed/21411619